CLINICAL TRIAL: NCT06848296
Title: Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of VSA012 Injection in Subjects with Paroxysmal Nocturnal Hemoglobinuria(PNH) Who Are Complement Inhibitor Naïve or Have Not Received Complement Inhibitor Therapy Recently
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of of VSA012 in Subjects with Paroxysmal Nocturnal Hemoglobinuria(PNH)
Acronym: VSA012-1001
Status: Not yet recruiting | Type: Observational
Sponsor: Visirna Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: VSA012-1002
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Weeks
Biospecimen Retention: Samples Without DNA — Blood Sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The complement system is an important component of the innate immune system. Abnormal activation, inadequate regulation and control of the complement system, as well as impaired and dysfunctional effector functions, underlie complement mediated diseases including PNH. VSA012 targeting complement system has the potential to treat a variety of diseases associated with abnormal activation of the complement system.The purpose of VSA012-1002 is to evaluate the safety, tolerability, pharmacokinetic, pharmacodynamics and efficacy of VSA012 Injection in subjects with PNH.

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, open-label Phase 1b study to evaluate the safety and tolerability, pharmacokinetic and pharmacodynamic profiles of VSA012 Injection in Chinese subjects with PNH, as well as to explore preliminary efficacy.

The VSA012 60 mg dose group and VSA012 120 mg dose group were initially proposed in this study; adjustments will be made based on data obtained in a single ascending dose study in healthy adult Chinese subjects (VSA012-1001) and stepwise data from this study, taking full account of subject safety. Enrollment in the 60 mg dose group of this study was not initiated until 15 days postdose safety assessments were completed for subjects in the 60 mg dose group of Study VSA012-1001; enrollment in the 120 mg dose group of Study VSA012-1001 was not initiated until 15 days postdose safety assessments were completed for subjects in the 120 mg dose group.

About 8 subjects with PNH will be enrolled in each group in this study and will receive VSA012 Injection 60 mg or V SA012 Injection 12 0 mg on D1 and D29, respectively; based on full consideration of the safety of subjects, the dosing regimen may be adjusted in combination with the data gradually obtained from the VSA012-1001 study and this study. Participants may receive concomitant supportive care permitted in this study throughout the study and continue to be followed for 24 weeks following completion of D29 dosing.

This study includes: Screening Period, Treatment Period, Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this clinical study, understand and follow study procedures and voluntarily sign the ICF;
* Body mass index (BMI) ≥ 18.0 kg/m2 , male or female, ≥ 18 years of age (including the critical value) at the time of signing the ICF;
* Confirmed diagnosis of PNH by clinical presentation and flow cytometry; flow cytometry within 6 months prior to or during screening consistent with granulocyte clonal size ≥ 10%;
* Hb < 100 g/L；
* Lactate dehydrogenase (LDH) > 1.5 × ULN；
* Subject is willing to receive 4-valent meningococcal vaccine, Streptococcus pneumoniae vaccine at least 14 days prior to dosing. If 4-valent meningococcal vaccine is administered within 3 years before the first dose, it may not be repeated; if S. pneumoniae vaccine is administered within 5 years, it may not be repeated;
* Agreed to use a highly effective method of contraception throughout the study and for 12 months after the last study dose.

Exclusion Criteria:

* History of hypersensitivity to VSA012 or its excipients;
* Use of any complement inhibitor within 3 months before screening or within 5 half-lives (whichever is longer);
* Infections prior to first dose;
* Prior splenectomy;
* Previously suspected/confirmed hereditary complement deficiency;
* History of recurrent invasive infection with encapsulated bacteria such as meningococcus or pneumococcus;
* Severe aplastic anemia (SAA) at screening and receiving immunosuppressive therapy;
* Patients with previous autoimmune diseases requiring systemic treatment, such as human immunodeficiency virus (HIV) infection, except for corticosteroid replacement therapy for thyroid, adrenal or pituitary insufficiency;
* History of allogeneic transplantation, stem cell transplantation, organ transplantation or other transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with PNH
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (AEs) and/or Serious Adverse Events (SAEs) | up to Day 196
preliminary efficacy | up to Day 196
  Percentage change from baseline in lactate dehydrogenase (LDH) by visit Change from baseline in hemoglobin (Hb) level by visit

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of VSA012 (First dose): Maximum Observed Plasma Concentration (Cmax) | Up to 48 hours post-dose
PK of VSA012(First dose): Time to Maximum Observed Plasma Concentration (Tmax) | Up to 48 hours post-dose
PK of VSA012(First dose)：Area under the concentration-time curve during the dosing interval (AUC 0-tau) | Up to 48 hours post-dose
PK of VSA012 (Multiple dose)：Trough concentration (C min) | Up to 48 hours post-dose
PK of VSA012 (Multiple dose)：Accumulation ratio of C max | Up to 48 hours post-dose
PK of VSA012 (Multiple dose)：AUC 0-tau | Up to 48 hours post-dose
PK of VSA012 (Multiple dose)：T max | Up to 48 hours post-dose
PK of VSA012 (Multiple dose)：C max (RacC max) | Up to 48 hours post-dose
PK of VSA012 (Multiple dose)：Accumulation ratio of AUC 0-tau (RacAUC 0-tau) | Up to 48 hours post-dose
Pharmacodynamic (PD) profile of VSA012:Change from baseline in complement factor B (CFB) and complement bypass pathway (CAP) activities | up to Day 196
PD of VSA012:Change from baseline in PNH clones, including number of PNH clones in erythrocytes, number of PNH clones in granulocytes, and number of PNH clones in monocytes | up to Day 196

IPD SHARING:
Plan to Share IPD: No